CLINICAL TRIAL: NCT00234065
Title: Post-marketing Study of Cilostazol: Study to Confirm Efficacy in Preventing Recurrent Cerebral Infarction in Comparison With Aspirin
Brief Title: Post-marketing Study of Cilostazol (Cilostazol Stroke Prevention Study 2)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Katsuhisa Saito, OPCJ
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: C02100-002; JapicCTI-050034; UMIN-CTR-C000000129
Record Dates: First submitted 2005-10-04; First posted 2005-10-06 (Estimated); Results first posted 2011-05-13 (Estimated); Last update posted 2011-06-10 (Estimated); Status verified 2011-06

CONDITIONS: Cerebral Infarction
MeSH Terms: conditions — Cerebral Infarction | interventions — Cilostazol; Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): cilostazol
  Interventions: Drug: Cilostazol
- 2 (Active Comparator): Aspirin
  Interventions: Drug: Aspirin

INTERVENTIONS:
Drug: Cilostazol — oral tablet, 100 mg twice a day and placebo of aspirin once a day, 1 to 5years
  Arms: 1
Drug: Aspirin — oral tablet, placebo of cilostazol twice a day and 81 mg once a day, 1 to 5 years
  Arms: 2

SUMMARY:
The purpose of this study is to investigate the efficacy of cilostazol in preventing recurrence of cerebral infarction and the safety of long-term administration of the drug (100 mg, twice daily) in patients with cerebral infarction (excluding cardiogenic cerebral embolism) in a multi-center, double-blind, parallel-group comparison with aspirin (81 mg, once daily).

ELIGIBILITY:
Inclusion Criteria:

1. Patients with stable medical conditions for 182 days (26 weeks) after occurrence of cerebral infarction
2. Patients in whom the infarct-related foci was detected by X-ray CT scan or MRI
3. Patients aged 20 to 80 years (inclusive) at time of consent
4. Patients with none of the following cardiac diseases that may be associated with cardiogenic cerebral embolism: mitral stenosis, prosthetic heart valve, endocarditis, myocardial infarction within 6 weeks after occurrence, ventricular aneurysm, endocardial thrombosis, mitral valve prolapse (patients less than 45 years of age in whom no other cause was identified), atrial fibrillation, sick sinus syndrome, idiopathic cardiomyopathy, and patent foramen ovale
5. Patients without asymptomatic cerebral infarction
6. Patients who have neither undergone nor are scheduled to undergo percutaneous transluminal angioplasty or revascularization for the treatment of cerebral infarction
7. Patients without severe disturbances/impairments following occurrence of cerebral

Exclusion Criteria:

1. Patients with hemorrhage or bleeding tendency (hemophilia, capillary fragility, intracranial hemorrhage, hemorrhage in the digestive tract, hemorrhage in the urinary tract, hemoptysis, and hemorrhage in the vitreous body)
2. Pregnant, possibly pregnant, or nursing women
3. Patients with ischemic heart failure
4. Patients with peptic ulcer
5. Patients with severer blood disorders
6. Patients with severe hepatic or renal
7. Patients with malignant neoplasm or patients who have received any therapy for malignant neoplasm within 5 years prior to entering the study
8. Patients with a history of hypersensitivity to salicylic acid formulations or ingredients of cilostazol tablets
9. Patients with aspirin asthma (asthma attacks induced by nonsteroidal antiinflammatory analgesic agents) or a history of aspirin asthma
10. Patients who are being treated with ticlopidine hydrochloride
11. Patients who are participating in another study for an investigational drug
12. Patients who are otherwise judged inappropriate for inclusion in the study by the investigators

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2800 (Actual)
Dates: Start 2003-12; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Masahiko Abe, Study Director — Division of New Product Evaluation and Development
Locations (1):
- Otsuka Pharmaceutical Co., Ltd., Tokyo, Japan

REFERENCES:
- [Result] Shinohara Y, Katayama Y, Uchiyama S, Yamaguchi T, Handa S, Matsuoka K, Ohashi Y, Tanahashi N, Yamamoto H, Genka C, Kitagawa Y, Kusuoka H, Nishimaru K, Tsushima M, Koretsune Y, Sawada T, Hamada C; CSPS 2 group. Cilostazol for prevention of secondary stroke (CSPS 2): an aspirin-controlled, double-blind, randomised non-inferiority trial. Lancet Neurol. 2010 Oct;9(10):959-68. doi: 10.1016/S1474-4422(10)70198-8. Epub 2010 Sep 15. PMID 20833591

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with non-cardioembolic ischemic stroke have been recruited at 278 study sites in Japan between December, 2003, and October, 2006.
Pre-assignment Details: No screening period
Groups:
- Cilostazol: cilostazol, oral tablet, 100 mg cilostazol
- Aspirin: Aspirin, oral tablet, 81 mg aspirin
Period: Overall Study
Arm/Group | Cilostazol | Aspirin
Started | 1356 | 1360
Completed | 881 | 1004
Not Completed | 475 | 356
Not completed — Adverse Event | 268 | 166
Not completed — Withdrawal by Subject | 73 | 56
Not completed — Physician Decision | 23 | 22
Not completed — Not Classified | 111 | 112

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cilostazol | Aspirin | Total
Number analyzed (Participants) | 1337 | 1335 | 2672
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 681 | 685 | 1366
  >=65 years | 656 | 650 | 1306
Age Continuous [Mean (Standard Deviation); unit: years] | 63.5 (9.2) | 63.4 (9.0) | 63.4 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 378 | 378 | 756
  Male | 959 | 957 | 1916
Region of Enrollment [Number; unit: participants]
  Japan | 1337 | 1335 | 2672

OUTCOME MEASURES:

1. Primary Outcome: Numbers of Patients With First Occurence of Stroke
Description: The endpoint in this measure is a composite endpoint of the first recurrence of cerebral infarction, or occurrence of cerebral haemorrhage or subarachnoid haemorrhage. The evaluation committee, whose members were unaware of patients' treatment assignment, adjudicated all trial endpoints.
Time Frame: From start of treatment to end of follow-up period ( follow-up periods : 29 months [Standard Deviation 16, range 1-59 months])
Population: Analyses were done using the full analysis set (FAS) of patients, as predetermined in the protocol. The full analysis set excluded patients who failed to satisfy inclusion criteria and those who violated exclusion criteria.
Measure: Number; unit: participants
Arm/Group | Cilostazol | Aspirin
Number analyzed (Participants) | 1337 | 1335
participants | 82 | 119
Statistical Analysis 1: Comparison: Cilostazol vs Aspirin; Statistical Analysis 1 for Number of Patients With First Occurrence of Stroke; Test type: Non-Inferiority or Equivalence — If the upper 95% CI limit for the HR of cilostazol to aspirin was 1.33 (4/3) or lower , cilostazol would be non-inferior to aspirin; p = 0.0357, Log Rank — The log-rank test was used to verify the superiority of CLZ to ASA only if non-inferiority was verified. The adjusted significance level for the superiority test of the endpoint was set at 0.0471 (two-tailed) according to the O'Brien-Fleming method; Hazard Ratio, log = 0.743, 95% CI 2-sided [0.564 to 0.981]

2. Secondary Outcome: Number of Patients With First Recurrence of Cerebral Infarction
Time Frame: From start of treatment to end of follow-up period (mean follow-up periods : 29 months [STANDARD DEVIATION 16, range 1-59 months])
Measure: Number; unit: participants
Arm/Group | Cilostazol | Aspirin
Number analyzed (Participants) | 1337 | 1335
participants | 72 | 88
Statistical Analysis 1: Comparison: Cilostazol vs Aspirin; Analyses were done using the full analysis set (FAS) of patients, as predetermined in the protocol. The full analysis set excluded patients who failed to satisfy inclusion criteria and those who violated exclusion criteria; Test type: Superiority or Other; p = 0.4189, Log Rank; Hazard Ratio, log = 0.88, 95% CI 2-sided [0.645 to 1.200]

3. Secondary Outcome: Number of Patients With First Occurrence of Ischaemic Cerebrovascular Disease
Description: The endpoint in this measure is a composite endpoint of the first recurrence of cerebral infarction or the first occurrence of transient ischaemic attack. The evaluation committee, whose members were unaware of patients' treatment assignment, adjudicated all trial endpoints.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Cilostazol | Aspirin
Number analyzed (Participants) | 1337 | 1335
participants | 86 | 103
Statistical Analysis 1: Comparison: Cilostazol vs Aspirin; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.4582, Log Rank; Hazard Ratio (HR) = 0.898, 95% CI 2-sided [0.675 to 1.194]

4. Secondary Outcome: Number of Deaths From Any Cause
Description: Number of deaths from any cause. The evaluation committee, whose members were unaware of patients' treatment assignment, adjudicated all trial endpoints.
Time Frame: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Cilostazol | Aspirin
Number analyzed (Participants) | 1337 | 1335
participants | 13 | 13
Statistical Analysis 1: Comparison: Cilostazol vs Aspirin; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.8600, Log Rank; Hazard Ratio (HR) = 1.072, 95% CI 2-sided [0.497 to 2.313]

5. Secondary Outcome: Number of Patients With First Occurrence of a Composite Endpoint of Stroke, Haemorrhagic Events, or Cardiovascular Events
Description: The endpoint in this measure is a composite endpoint of the first recurrence of cerebral infarction, or occurrence of cerebral haemorrhage, subarachnoid haemorrhage, transient ischaemic attack, angina pectris, myocardial infarction, heart failure, or haemorrhage requiring hospital admission. The evaluation committee, whose members were unaware of patients' treatment assignment, adjudicated all trial endpoints.
Time Frame: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Cilostazol | Aspirin
Number analyzed (Participants) | 1337 | 1335
participants | 138 | 186
Statistical Analysis 1: Comparison: Cilostazol vs Aspirin; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0437, Log Rank; Hazard Ratio (HR) = 0.799, 95% CI 2-sided [0.643 to 0.994]

6. Other Pre Specified Outcome: Number of Patients With First Occurrence of Haemorrhagic Event
Description: The endpoint in this measure is a composite endpoint of the first occurrence of cerebral haemorrhage, subarachnoid haemorrhage or haemorrhage requiring hospital admission. The evaluation committee, whose members were unaware of patients' treatment assignment, adjudicated all trial endpoints.
Time Frame: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Cilostazol | Aspirin
Number analyzed (Participants) | 1337 | 1335
participants | 23 | 57
Statistical Analysis 1: Comparison: Cilostazol vs Aspirin; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0004, Log Rank; Hazard Ratio (HR) = 0.458, 95% CI 2-sided [0.296 to 0.711]

ADVERSE EVENTS:
Time Frame: From start of treatment to end of follow-up period (mean follow-up periods : 29 months [STANDARD DEVIATION 16, range 1-59 months])
Arm/Group | Cilostazol | Aspirin
Serious Adverse Events (participants affected / at risk) | 372/1337 | 433/1335
Other Adverse Events (participants affected / at risk) | 1267/1337 | 1260/1335
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cilostazol (N=1337) | Aspirin (N=1335)
Anaemia (Blood and lymphatic system disorders) | 2 | 5
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Anaemia macrocytic (Blood and lymphatic system disorders) | 0 | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 2
Hypochromic anaemia (Blood and lymphatic system disorders) | 0 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 4
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 10 | 3
Angina pectoris (Cardiac disorders) | 7 | 6
Atrial fibrillation (Cardiac disorders) | 6 | 0
Acute myocardial infarction (Cardiac disorders) | 4 | 7
Cardiac failure (Cardiac disorders) | 3 | 4
Cardiac failure congestive (Cardiac disorders) | 3 | 1
Angina unstable (Cardiac disorders) | 2 | 4
Cardiac failure acute (Cardiac disorders) | 2 | 2
Ventricular extrasystoles (Cardiac disorders) | 2 | 1
Myocardial ischaemia (Cardiac disorders) | 1 | 3
Prinzmetal angina (Cardiac disorders) | 1 | 1
Intracardiac thrombus (Cardiac disorders) | 1 | 0
Stress cardiomyopathy (Cardiac disorders) | 1 | 0
Aortic valve stenosis (Cardiac disorders) | 0 | 1
Atrial flutter (Cardiac disorders) | 0 | 2
Atrioventricular block complete (Cardiac disorders) | 0 | 1
Atrioventricular block second degree (Cardiac disorders) | 0 | 1
Coronary artery stenosis (Cardiac disorders) | 0 | 3
Silent myocardial infarction (Cardiac disorders) | 0 | 1
Hydrocele (Congenital, familial and genetic disorders) | 1 | 0
Intestinal malrotation (Congenital, familial and genetic disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 4 | 1
Vertigo positional (Ear and labyrinth disorders) | 3 | 2
Sudden hearing loss (Ear and labyrinth disorders) | 3 | 3
Meniere's disease (Ear and labyrinth disorders) | 1 | 0
Vertigo labyrinthine (Ear and labyrinth disorders) | 1 | 2
Cataract (Eye disorders) | 22 | 17
Macular oedema (Eye disorders) | 2 | 0
Cataract subcapsular (Eye disorders) | 1 | 0
Diabetic retinal oedema (Eye disorders) | 1 | 0
Pterygium (Eye disorders) | 1 | 1
Vitreous haemorrhage (Eye disorders) | 1 | 1
Entropion (Eye disorders) | 1 | 0
Ulcerative keratitis (Eye disorders) | 1 | 0
Amaurosis (Eye disorders) | 0 | 1
Cataract diabetic (Eye disorders) | 0 | 1
Diabetic retinopathy (Eye disorders) | 0 | 1
Macular degeneration (Eye disorders) | 0 | 1
Retinal detachment (Eye disorders) | 0 | 1
Retinal haemorrhage (Eye disorders) | 0 | 1
Retinal vein occlusion (Eye disorders) | 0 | 1
Macular hole (Eye disorders) | 0 | 2
Tolosa-Hunt syndrome (Eye disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 11 | 5
Colonic polyp (Gastrointestinal disorders) | 10 | 7
Gastric ulcer (Gastrointestinal disorders) | 6 | 4
Enterocolitis (Gastrointestinal disorders) | 2 | 2
Haemorrhoids (Gastrointestinal disorders) | 2 | 3
Hiatus hernia (Gastrointestinal disorders) | 2 | 0
Intestinal obstruction (Gastrointestinal disorders) | 2 | 1
Periodontitis (Gastrointestinal disorders) | 2 | 3
Reflux oesophagitis (Gastrointestinal disorders) | 2 | 0
Anal fistula (Gastrointestinal disorders) | 1 | 0
Colitis ischaemic (Gastrointestinal disorders) | 1 | 4
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1 | 1
Gastric polyps (Gastrointestinal disorders) | 1 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 | 9
Gastrointestinal disorder (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 4
Ileus (Gastrointestinal disorders) | 1 | 2
Ileus paralytic (Gastrointestinal disorders) | 1 | 0
Mallory-Weiss syndrome (Gastrointestinal disorders) | 1 | 0
Melaena (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Peritonitis (Gastrointestinal disorders) | 1 | 0
Large intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Diverticulitis intestinal haemorrhagic (Gastrointestinal disorders) | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Food poisoning (General disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Gastritis erosive (Gastrointestinal disorders) | 0 | 1
Gastroduodenal ulcer (Gastrointestinal disorders) | 0 | 2
Gingival hyperplasia (Gastrointestinal disorders) | 0 | 1
Large intestinal ulcer (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Varices oesophageal (Gastrointestinal disorders) | 0 | 1
Disuse syndrome (General disorders) | 3 | 1
Granuloma (Gastrointestinal disorders) | 2 | 0
Sudden death (General disorders) | 2 | 2
Chest pain (General disorders) | 1 | 1
Mass (General disorders) | 1 | 0
Cardiac death (General disorders) | 1 | 0
Gait disturbance (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 5 | 3
Bile duct stone (Hepatobiliary disorders) | 3 | 2
Cholangitis (Hepatobiliary disorders) | 2 | 0
Autoimmune hepatitis (Hepatobiliary disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 3
Liver disorder (Hepatobiliary disorders) | 1 | 1
Biliary cirrhosis primary (Hepatobiliary disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 2
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 1
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 1
Pneumonia (Infections and infestations) | 8 | 9
Gastroenteritis (Infections and infestations) | 5 | 3
Appendicitis (Infections and infestations) | 3 | 1
Bronchitis (Infections and infestations) | 3 | 1
Herpes zoster (Infections and infestations) | 3 | 1
Pyelonephritis (Infections and infestations) | 3 | 3
Pyelonephritis acute (Infections and infestations) | 3 | 3
Sinusitis (Infections and infestations) | 2 | 0
Urinary tract infection (Infections and infestations) | 2 | 3
Enteritis infectious (Infections and infestations) | 2 | 0
Appendicitis perforated (Infections and infestations) | 1 | 0
Bronchopneumonia (Infections and infestations) | 1 | 2
Cellulitis (Infections and infestations) | 1 | 3
Diverticulitis (Infections and infestations) | 1 | 0
Herpes virus infection (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 1
Nasopharyngitis (Infections and infestations) | 1 | 1
Postoperative wound infection (Infections and infestations) | 1 | 0
Retroperitoneal abscess (Infections and infestations) | 1 | 0
Viral infection (Infections and infestations) | 1 | 1
Anal abscess (Infections and infestations) | 1 | 2
Postoperative abscess (Infections and infestations) | 1 | 0
Extradural abscess (Infections and infestations) | 1 | 0
Osteomyelitis (Infections and infestations) | 0 | 1
Pelvic abscess (Infections and infestations) | 0 | 1
Pseudomembranous colitis (Infections and infestations) | 0 | 1
Varicella (Infections and infestations) | 0 | 1
Anogenital warts (Infections and infestations) | 0 | 1
Pneumonia bacterial (Infections and infestations) | 0 | 1
Pneumocystis jiroveci pneumonia (Infections and infestations) | 0 | 1
Enterocolitis bacterial (Infections and infestations) | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 6 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 6 | 4
Contusion (Injury, poisoning and procedural complications) | 6 | 2
Subdural haematoma (Injury, poisoning and procedural complications) | 3 | 2
Facial bones fracture (Injury, poisoning and procedural complications) | 2 | 0
Hand fracture (Injury, poisoning and procedural complications) | 2 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 2 | 0
Rib fracture (Injury, poisoning and procedural complications) | 2 | 4
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 1
Carbon monoxide poisoning (Injury, poisoning and procedural complications) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Injury (Injury, poisoning and procedural complications) | 1 | 0
Multiple fractures (Injury, poisoning and procedural complications) | 1 | 0
Spinal cord injury (Injury, poisoning and procedural complications) | 1 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 1
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 | 2
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Muscle strain (Infections and infestations) | 1 | 1
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0
Eye injury (Injury, poisoning and procedural complications) | 1 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Renal injury (Injury, poisoning and procedural complications) | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Burns third degree (Injury, poisoning and procedural complications) | 0 | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 2
Compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Extradural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 0 | 2
Forearm fracture (Injury, poisoning and procedural complications) | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1
Joint sprain (Injury, poisoning and procedural complications) | 0 | 1
Open fracture (Injury, poisoning and procedural complications) | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 2
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1
Brain contusion (Injury, poisoning and procedural complications) | 0 | 2
Meniscus lesion (Injury, poisoning and procedural complications) | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1
Skull fracture (Injury, poisoning and procedural complications) | 0 | 2
Limb traumatic amputation (Injury, poisoning and procedural complications) | 0 | 1
Blood urea increased (Investigations) | 2 | 1
Blood glucose increased (Investigations) | 1 | 0
Blood pressure increased (Investigations) | 1 | 1
Blood glucose fluctuation (Investigations) | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 1
Blood potassium increased (Investigations) | 0 | 1
Platelet count decreased (Investigations) | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 5 | 6
Hypoglycaemia (Metabolism and nutrition disorders) | 5 | 1
Anorexia (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 2
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Back pain (Metabolism and nutrition disorders) | 3 | 3
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 2
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 1
Spinal ligament ossification (Musculoskeletal and connective tissue disorders) | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 2
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Periostitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Axillary mass (Musculoskeletal and connective tissue disorders) | 0 | 1
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 2
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 | 8
Large intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 | 4
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 4
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Bladder papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Carcinoid tumour of the gastrointestinal tract (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant neoplasm of renal pelvis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Small intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Gastric adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 4
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Spinal cord neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Adenoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Haemangioma of liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Kaposi's sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Liposarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Small cell lung cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ureteric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Salivary gland adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pancreatic carcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Adrenal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastatic gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebral infarction (Nervous system disorders) | 62 | 84
Transient ischaemic attack (Nervous system disorders) | 8 | 9
Dizziness (Nervous system disorders) | 7 | 6
Cerebral haemorrhage (Nervous system disorders) | 4 | 25
Epilepsy (Nervous system disorders) | 3 | 3
Loss of consciousness (Nervous system disorders) | 3 | 1
Facial palsy (Nervous system disorders) | 2 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 2 | 4
Syncope (Nervous system disorders) | 2 | 2
Convulsion (Nervous system disorders) | 1 | 3
Dementia Alzheimer's type (Nervous system disorders) | 1 | 0
Haemorrhagic cerebral infarction (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 1
Hypoglycaemic coma (Nervous system disorders) | 1 | 0
Intraventricular haemorrhage (Nervous system disorders) | 1 | 0
Paralysis (Nervous system disorders) | 1 | 0
Presenile dementia (Nervous system disorders) | 1 | 0
Ruptured cerebral aneurysm (Nervous system disorders) | 1 | 0
Vertebral artery stenosis (Nervous system disorders) | 1 | 1
Reversible ischaemic neurological deficit (Nervous system disorders) | 1 | 0
Thalamus haemorrhage (Nervous system disorders) | 1 | 1
Putamen haemorrhage (Nervous system disorders) | 1 | 0
Thrombotic cerebral infarction (Nervous system disorders) | 1 | 1
Amyotrophic lateral sclerosis (Nervous system disorders) | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 0 | 1
Cerebellar haemorrhage (Nervous system disorders) | 0 | 1
Cervicobrachial syndrome (Nervous system disorders) | 0 | 1
Dysarthria (Nervous system disorders) | 0 | 1
Myelopathy (Nervous system disorders) | 0 | 1
Petit mal epilepsy (Nervous system disorders) | 0 | 1
Sciatica (Nervous system disorders) | 0 | 1
Vertebral artery occlusion (Nervous system disorders) | 0 | 1
Delirium (Psychiatric disorders) | 2 | 0
Anxiety disorder (Psychiatric disorders) | 2 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Completed suicide (Psychiatric disorders) | 1 | 2
Suicide attempt (Psychiatric disorders) | 1 | 3
Alcoholism (Psychiatric disorders) | 0 | 2
Depression (Psychiatric disorders) | 0 | 1
Dissociative disorder (Psychiatric disorders) | 0 | 1
Mania (Psychiatric disorders) | 0 | 1
Adjustment disorder (Psychiatric disorders) | 0 | 1
Calculus bladder (Renal and urinary disorders) | 2 | 0
Calculus ureteric (Renal and urinary disorders) | 1 | 4
Calculus urethral (Renal and urinary disorders) | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 2
Nephrolithiasis (Renal and urinary disorders) | 1 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 1
Bladder prolapse (Renal and urinary disorders) | 1 | 0
Acute prerenal failure (Renal and urinary disorders) | 0 | 1
Calculus urinary (Renal and urinary disorders) | 0 | 1
Glomerulonephritis rapidly progressive (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 2
Nephritis (Renal and urinary disorders) | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1
Renal impairment (Renal and urinary disorders) | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 1
Uterine prolapse (Reproductive system and breast disorders) | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 0 | 2
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Diaphragmatic disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Status asthmaticus (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 0
Neurodermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Hypoaesthesia facial (Skin and subcutaneous tissue disorders) | 0 | 1
Skin mass (Skin and subcutaneous tissue disorders) | 0 | 1
Shock haemorrhagic (Vascular disorders) | 2 | 0
Aneurysm (Vascular disorders) | 1 | 0
Aortic aneurysm (Vascular disorders) | 1 | 1
Aortic aneurysm rupture (Vascular disorders) | 1 | 0
Varicose vein (Vascular disorders) | 1 | 3
Arteriosclerosis obliterans (Vascular disorders) | 1 | 0
Peripheral artery aneurysm (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cilostazol (N=1337) | Aspirin (N=1335)
Palpitations (Cardiac disorders) | 156 | 71
Tachycardia (Cardiac disorders) | 89 | 21
Diarrhoea (Gastrointestinal disorders) | 164 | 85
Constipation (Gastrointestinal disorders) | 110 | 155
Dental caries (Gastrointestinal disorders) | 93 | 114
Periodontitis (Gastrointestinal disorders) | 77 | 64
Nasopharyngitis (Infections and infestations) | 546 | 590
Contusion (Injury, poisoning and procedural complications) | 128 | 121
Blood glucose increased (Investigations) | 92 | 79
Blood pressure increased (Investigations) | 71 | 88
Blood creatine phosphokinase increased (Investigations) | 67 | 76
Diabetes mellitus (Metabolism and nutrition disorders) | 96 | 75
Back pain (Musculoskeletal and connective tissue disorders) | 160 | 165
Arthralgia (Musculoskeletal and connective tissue disorders) | 118 | 102
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 73 | 55
Headache (Nervous system disorders) | 312 | 217
Dizziness (Nervous system disorders) | 124 | 92
Insomnia (Psychiatric disorders) | 81 | 96
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 97 | 105
Eczema (Skin and subcutaneous tissue disorders) | 97 | 104
Hypertension (Vascular disorders) | 120 | 185

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No